CLINICAL TRIAL: NCT01540188
Title: Development of a Family Intervention to Address Drug Use and HIV in Vietnam
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Principal Investigator, Li Li, Principal investigator, Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34DA029493 (NIH)
Record Dates: First submitted 2012-02-09; First posted 2012-02-28 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Quality of Life
Keywords: Drug user; Family member; Intervention; Community; Support
MeSH Terms: conditions — Drug Misuse | interventions — Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Starndard care arm (No Intervention): Participants of the standard care arm are control groups of IDUs and family members. They do not attend intervention sessions.
- Intervention arm (Experimental): Intervention for IDUs: there are 4 sessions of the intervention with the following titles: My family, my health, my actions, my community.
  Intervention for family members: there are 4 intervention sessions for family members covering the following topics: my family, my responsibility, my support and my community
  Interventions: Behavioral: Family Intervention to Address Drug Use and HIV in Vietnam

INTERVENTIONS:
Behavioral: Family Intervention to Address Drug Use and HIV in Vietnam — Intervention for IDUs: there are 4 sessions of the intervention with the following titles: My family, my health, my actions, my community.
  Intervention for family members: there are 4 intervention sessions for family members covering the following topics: my family, my responsibility, my support and my community
  Arms: Intervention arm

SUMMARY:
Vietnam is currently experiencing two epidemics -- injection drug use and HIV. HIV infection is rising rapidly, primarily among injecting drug users (IDUs). Most young IDUs keep daily contact with their family or live in their parent's home. The burden on their families is substantial, and even greater if the IDU is HIV+. In this study, the investigators conduct an intervention pilot to develop and evaluate a family intervention to improve outcomes over time for Vietnamese IDUs and their families. This two-year study is conducted in Phu Tho, a province located about 80 km from Hanoi, Vietnam's capital.

Two teams with complementary expertise collaborate to implement this study: the UCLA team and the Vietnamese team from the Vietnam National Institute of Hygiene & Epidemiology (NIHE). The study has two phases:

* In Phase 1, the investigators develop the content, format and an implementation plan for the intervention from a focus group of 10 service providers, administrators and community leaders, and through in-depth interviews with 40 IDUs (20 HIV+ and 20 HIV-) recruited from the local drug rehabilitation center (the "06 Center") and from two local communities (Duu Lau and Gia Cam), as well as in-depth interviews with 20 of the IDUs family members (FM). Based on the findings, the investigators collaborate on designing a Vietnamese-specific family intervention for IDUs and their family members.
* In Phase 2, the investigators pilot the intervention in the local commune health centers in Viet Tri, Phu Tho. Eighty IDUs (HIV+/HIV-) and 80 of their family members are recruited from 4 communes and the 06 Center in Viet Tri city, and randomized into a intervention group and a control group. After the 4-week intervention, 3-month and 6-month follow-ups are conducted to assess the effectiveness of the intervention. Participants randomized to the control group only complete the assessments (baseline, 3-, and 6-month) at the same time points.

DETAILED DESCRIPTION:
Vietnam is facing the challenge of dual epidemics -injection drug use and HIV. HIV infection is rising exponentially, primarily among injecting drug users (IDUs). Because Vietnamese are highly family oriented, most young IDUs have daily family contact or live in their parents' homes. The burden on the family is substantial, and even greater if the IDU is HIV+. The investigators hypothesize that with assistance, families can be part of the solution for both HIV and HIV+ IDU. This family intervention in Vietnam is based on the Social Action Theory and Social Network Theory, aimed at increasing families' capacities to effectively cope with the impact of IDUs and HIV. The study provides an opportunity to test culturally-specific intervention content and delivery. In addition, the intervention pilot will provide an opportunity to obtain project implementation experience in the local settings. The study also provides the opportunity to pilot test outcome measures.

The specific aims of the study are:

1. To document the challenges of drug use and HIV for IDUs and their family members;
2. To examine the acceptability and feasibility of a family-based intervention for IDU and their family members;
3. To examine whether the IDUs and family members in the intervention group, compared to those in the standard care group, will have significantly improved health, mental health, and quality of life outcomes, including health seeking, reduced sexual and drug use risk behaviors, increased HIV testing, and reduced caregiver burden; and
4. To examine how outcomes of the IDUs and family members are mediated by family indicators such as family cohesion, stress and symptom management, stigma and harm reduction, HIV disclosure, and treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* IDUs:

  * Age 18 or over
  * Either HIV + or HIV- in blood test
  * A current or past injection drug user
  * Disclosure of drug use status and HIV positive status (if positive) to their family members
  * Voluntary informed consent

Family members:

* Age 18 or over
* Immediate or extended family member of an IDU and living with the IDU.
* Previous knowledge of the drug use and HIV status (if positive) of the IDU.
* Voluntary informed consent

Exclusion Criteria:

* IDUs :

  * Inability to give informed consent
  * Has not disclosed the drug use status and HIV status (if positive) to family member
  * Not a current or past injection drug user

Family members:

* Inability to give informed consent
* Does not know the drug use status and HIV status (if positive) of the IDU in their family

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Physical health | Changes from baseline to 3- and 6-month follow-up
  The IDUs will be assessed using the Medical Outcomes Study (MOS) Short-Form 36 (SF-36). The MOS-SF-36 consists of the following domains: physical functioning; role limitation (physical); role limitation (emotional); social functioning; mental health; energy/vitality; pain; and general health perception. The score for each domain ranges from 0 to 100 with higher values indicating higher functional status.
Mental health | Changes from baseline to 3- and 6-month follow-up
  All of the participants including both IDUs and family members will be assessed by the Zung Self-Rating Depression Scale. This measure, developed by the World Health Organization, is a 20-item self-report scale that is widely used as a screening tool, covering affective, psychological and somatic symptoms associated with depression. Results from this measure will be used as an indicator of psychological (including psychosis) and emotional functioning that can be associated with drug use.

SECONDARY OUTCOMES:
Drug use | Changes from baseline to 3- and 6-month follow-up
  Measures will include data on alcohol use and other drug use. For the IDU participants, their drug use will be measured by a biomarker (Urine drug screen) at the baseline, since the drug rehabilitation sites routinely collect urine to test for drug use. Positive results will be interpreted as signifying drug use, regardless of self-report.
Sexual risk | Changes from baseline to 3- and 6-month follow-up
  This is assessed using the Risk Assessment Battery (RAB; Metzger, 1995) Collecting data on self-reported HIV risk behaviors is especially relevant as there is a well-documented association between drug use and participation in high risk sexual behaviors related to HIV-transmission.
Caregiver burden | Changes from baseline to 3- and 6-month follow-up
  This is assessed using the Perceived Caregiver Burden Scale (PCB) (Stommel et al., 1990). This scale has been used in our studies in Thailand and China (Lee et al., 2009b) to assess caregiver burden in terms of perceptions and feelings about family members' physical and emotional health, family relationships, social life, work, and finances.
Family/social support | Changes from baseline to 3- and 6-month follow-up
  This is measured by two instruments. Social Support Questionnaire (Short; SSQ6) is a 6-item assessment to measure satisfaction of social support. Number of social support providers is captured up to 9 people in various support dimensions (Sarason et al., 1983). Medical Outcomes Study- Social Support Scale (MOS-SS) is a 20-item scale that measures the strength of perceived social support available. The scale consists of five dimensions: emotional support, informational support, tangible support, positive social interaction, and affection.

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, Ph.D, Principal Investigator — University of California, Los Angeles
Locations (1):
- Commune health centers, Việt Trì, Phu Tho, Vietnam